CLINICAL TRIAL: NCT07175142
Title: Assessment of Psychological Distress, Sleep Quality, and Halitosis in Patients With Obesity: Protocol for an Observational Study in the Preoperative Period of Bariatric Surgery
Brief Title: Halitosis, Sleep and Mental Health in Bariatric Surgery Candidates
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nove de Julho (Other)
Collaborators: Universidade Metropolitana de Santos (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Other Study IDs: HalitosisBariatricStudy
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Bariatric Surgery Candidate; Halitosis; Sleep Disorder; Stress, Psychological
MeSH Terms: conditions — Obesity; Halitosis; Sleep Wake Disorders; Stress, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate psychological distress, sleep quality, and halitosis in obese patients during the preoperative period of bariatric surgery. A total of 110 adults will be assessed using validated questionnaires and a portable halitosis detector. The results may contribute to improving strategies for comprehensive care in this population.

DETAILED DESCRIPTION:
This is an observational, cross-sectional study designed to assess the prevalence of psychological distress, sleep quality, and halitosis in obese patients who are candidates for bariatric surgery in the metropolitan region of Santos, Brazil. Participants (n=110) will be recruited during the preoperative assessment period at the Interprofessional Outpatient Clinic of Universidade Metropolitana de Santos (UNIMES).

Psychological distress will be measured using the Depression, Anxiety, and Stress Scale (DASS-21). Sleep quality will be evaluated with the Pittsburgh Sleep Quality Index (PSQI-BR). Halitosis will be assessed by clinical anamnesis, lingual coating index, and a KKCare Portable Detector.

The main outcomes are the prevalence of stress, anxiety, and depression; the prevalence of poor sleep quality; and the prevalence of halitosis in this patient population. The study will also investigate possible associations between these psychosocial and oral health variables. Data will be analyzed using descriptive statistics and binary logistic regression.

The findings are expected to support strategies to improve multidisciplinary care and enhance the quality of life of obese patients preparing for bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with a diagnosis of obesity
* Referred for psychological care at the "Rosinha Viegas" Interprofessional Outpatient Clinic during preoperative preparation for bariatric surgery (Brazilian public health system - SUS)

Exclusion Criteria:

* Individuals with cognitive or neurological limitations that impair understanding or participation in the assessment procedures

Individuals who refuse or withdraw consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adult patients in the metropolitan region of Santos, Brazil, who are undergoing multidisciplinary assessment in preparation for bariatric surgery within the Brazilian public health system (SUS).
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of psychological distress (stress, anxiety, and depression) | Baseline
  Psychological distress will be measured using the Depression, Anxiety, and Stress Scale - short form (DASS-21), validated for Portuguese. The scale consists of 21 items equally distributed among depression, anxiety, and stress domains. Scores will be classified according to standardized cutoff points.

SECONDARY OUTCOMES:
Prevalence of halitosis in obese patients before bariatric surgery | Baseline
  Halitosis will be evaluated by clinical anamnesis, lingual coating index, and KKCare Portable Detector, which measures volatile sulfur compounds and provides classification across five levels of halitosis severity.